CLINICAL TRIAL: NCT06185959
Title: Examining the Feasibility and Impact of a Novel Psychoeducation and Process Group for Asian and Asian American Psychiatric Outpatients
Brief Title: Evaluating a New Mental Health Group for Asians and Asian Americans
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lisa Zhang, Clinical Assistant Professor, Stanford University
Other Study IDs: 72936
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in a Psychoeducation and Process Group for Asian and Asian American Psychiatric Outpatients
  Interventions: Behavioral: Psychoeducation and Process Group for Asian and Asian American Psychiatric Outpatients

INTERVENTIONS:
Behavioral: Psychoeducation and Process Group for Asian and Asian American Psychiatric Outpatients — Participants will be individuals enrolling in a 1.5 hour weekly therapy group lasting 12 weeks and will be invited to participate in research on group processes and outcomes. The psychoeducation and process group will be a 12-session weekly closed group with 10-15 participants per group (2-3 groups total) conducted via Zoom to enhance accessibility and reduce barriers to care. Groups will be co-led by licensed clinical psychologists with experience providing both group psychotherapy and culturally responsive services. Group sessions will include brief check-ins, collaborative agenda-setting, a mini-didactic, individual reflection, and group discussion. The didactics curriculum will include topics such as intergenerational trauma, cultural differences in emotional expression, the model minority myth, family dynamics, racism, and positive connections to culture.

SUMMARY:
This study's overarching aim is to evaluate a new psychoeducation and process group for Asian and Asian American psychiatric outpatients. This is a 12 week mental health group which will focus on both educational content related to Asian mental health as well as increasing connection between group members. We hypothesize that participants in the group will experience a decrease in psychiatric symptoms at the conclusion of the group compared to their symptoms at the beginning of group. We also hypothesize that participants will feel more socially connected after the group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Participants must identify as Asian or Asian American
* Sufficient English proficiency to participate in a psychotherapy group conducted in English

Exclusion Criteria:

* Unable to provide written informed consent
* Elevated suicide risk (e.g. recent active suicidal ideation, past-year suicide attempt) without a current individual mental health provider
* Any other challenges that would preclude participation in group psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age range is 18 years and older. All genders are eligible. For ethnic background, to be eligible for this study, participants must identify as Asian or Asian American due to the group under investigation being specifically designed as an Asian and Asian American Psychoeducation and Process Group.
  The research study will be offered to all patients enrolling in the Asian and Asian American Psychoeducation and Process Group in the Stanford Department of Psychiatry & Behavioral Sciences. The purpose of this study is to evaluate patient experiences in this psychoeducation and process group, so participants will be limited to those enrolling in the group as part of their clinical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Once at baseline, once at 6 weeks, once at 12 weeks
  Depression symptoms assessed on 4-point Likert scale. Score range from 0 to 27, with higher scores representing more severe depression symptoms
Generalized Anxiety Disorder Screener-7 (GAD-7) | Once at baseline, once at 6 weeks, once at 12 weeks
  Anxiety symptoms assessed on 4-point Likert scale. Score range from 0 to 21, with higher scores representing more severe anxiety symptoms

SECONDARY OUTCOMES:
Social Connectedness Scale | Once at baseline, once at 12 weeks
  Subjective social connectedness assessed on 6-point Likert scale. Score range from 20 to 120, with higher scores representing higher perceived social connectedness
Rosenberg Self-Esteem Scale | Once at baseline, once at 12 weeks
  Subjective self-esteem assessed on 4-point Likert scale. Score range from 10 to 40, with higher scores representing higher self-esteem
Self-Stigma of Seeking Help Scale | Once at baseline, once at 12 weeks
  Help-seeking self-stigma assessed on 5-point Likert scale. Score range from 10 to 50, with higher scores representing higher self-stigma of seeking help

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zhang, PhD, Principal Investigator — Stanford University; Melanie Hom, PhD, Principal Investigator — Stanford University; Stacy Lin, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University - Department of Psychiatry and Behavioral Sciences, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No